CLINICAL TRIAL: NCT02905760
Title: Efficacy of Furosemide Versus Vascular Filling in Patients With Acute Myocardial Infarction With Right Ventricular Extension: A Multicentric Randomized Controlled Trial
Brief Title: Efficacy of Furosemide Versus Vascular Filling in Patients With Acute Myocardial Infarction
Acronym: FAMIE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P150801
Record Dates: First submitted 2016-07-31; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myocardial Infarction With Right Ventricular Extension
Keywords: Acute Myocardial Infarction; Right ventricular infarction; Diuretic; Fluid Expansion
MeSH Terms: interventions — Furosemide; Diuretics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Furosemide (Experimental): Furosemide and Placebo filling (Glucose 5%).
  Interventions: Drug: Furosemide; Drug: Placebo filling
- Fluid expansion (Active Comparator): Placebo furosemide (Glucose 5%) and Vascular filling
  The vascular filling is the gold standard in the treatment of acute myocardial infarction
  Interventions: Drug: Placebo furosemide; Drug: Vascular filling

INTERVENTIONS:
Drug: Furosemide — Furosemide: Special LASILIX (250 mg/25 ml) solution for injection reconditioned glass bottle like "penicillin" of 80mg/8mL. Injection by slow intravenous (1 to 2 minutes per 80mg vial)
  Other Names: Diuretics, LASILIX.
  Arms: Furosemide
Drug: Placebo filling — Placebo filling: Glucose 5%, 500mL infused over 30 minutes.
  Other Names: G5
  Arms: Furosemide
Drug: Placebo furosemide — Placebo furosemide: glucose 5% for injection reconditioned glass bottle like "penicillin" of 80mg/8mL. Injection by slow intravenous (1 to 2 minutes per 80mg vial).
  Other Names: G5
  Arms: Fluid expansion
Drug: Vascular filling — Vascular filling: Sodium 0.9% 500mL infused over 30 minutes.
  Other Names: Fluid expansion, Sodium Chloride NaCl 0.9%.
  Arms: Fluid expansion

SUMMARY:
Right ventricular necrosis increases patient in hospital mortality and can be observed in 20-50% of patients admitted for during acute myocardial infarction. Current guidelines recommend managing cardiogenic shock related to right ventricular necrosis by optimizing RV load using fluid expansion and if insufficient adding inotropic support. However, several experimental studies reported a potential deleterious effect of right ventricular dilation related to fluid expansion because right and left ventricular interaction decreases stroke volume and cardiac output. Consistently with these finding, a study on a small patient sample conducted at Henri Mondor Hospital demonstrates the safety and efficiency of furosemide in patients with right ventricular necrosis.

The present study is a phase 3, interventional, prospective, randomized, multicenter, double-blind analysis by intention to treat.

The main objective is to demonstrate improved hemodynamic parameters in the short term in patients admitted for acute myocardial infarction with extension RV treated with furosemide.

The primary endpoint is compare the change in cardiac output in patients admitted and treated by either fluid expansion or furosemide.

The study population will consist in 88 patients and the duration of subjects' participation will be one month.

ELIGIBILITY:
Inclusion Criteria

* Age >18 years
* Inferior acute myocardial infarction (≤J + 7)
* Right ventricular extension defined by one following echocardiographic criteria:

  * Dilatation of the right ventricle (RV/LV area> 0.9)
  * RV dysfunction defined by TAPSE <16mm or S velocity <10cm.s-1
  * Akinesia or hypokinesia of two contiguous segments of the right ventricle
  * Decrease of pitch on lung failure flow <150ms
* Inferior vena cava dilatation (≥20mm) and non-compliant (changes <50%) associated with one hemodynamic instability criteria:

  * Oliguria (diuresis <800mL/24h or 0.5mL/kg/min)
  * Systolic blood pressure <100mmHg
  * Oxygen saturation <91% on room air
  * Bradycardia (heart rate <60/min, not valid for patients on beta-blockers).
* Informed consent for study participation signed.

Exclusion Criteria

* Minor and pregnant woman
* Mechanical complications of myocardial infarct
* Patients who received> 40mg diuretic /day during the last 15 days
* Hypersensitivity to furosemide or any of its excipients
* Aortic stenosis (area <1 cm² or mean gradient> 40mmHg), mitral or aortic regurgitation grade ≥3
* Catecholamine support for left ventricular failure with left ventricular ejection fraction <35%
* Renal impairment defined by a serum creatinine> 200μmol / mL
* Sodium and water retention
* Urinary tract obstruction
* Hypovolemia or dehydration
* Severe hypokalemia (K + <3 mmol / L)
* Severe hyponatremia (Na + <125 mmol / L)
* Hepatitis ongoing, liver failure or hepatic encephalopathy
* No affiliation to a social security scheme or other social protection scheme
* Private Patient of liberty or under legal protection (guardianship)
* Inability or refusal to understand or refusal to sign the informed consent from study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-11 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in cardiac output (measured by Doppler method) defined by an increase of more than 10% 24 hours after administration of the treatment in patients admitted and treated by either fluid expansion or furosemide. | At Hour 24

SECONDARY OUTCOMES:
Intra-hospital mortality | an average of 10 days after inclusion
Rate of inotropic support | an average of 10 days after inclusion
Number of hemodynamic instability requiring fluid expansion | an average of 10 days after inclusion
Change in systolic blood | Hour 24
Change in heart rate | Hour 24
Urine output | Hour 24
The duration of hospitalization in intensive care | an average of month 1
Hospitalizations for cardiovascular reason one month after acute myocardial infarction | month 1
One month mortality | month 1

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Lim, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No